CLINICAL TRIAL: NCT07055815
Title: Impact of Digital Screen Time in Progression of Myopia in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/831
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Progression of Myopia — The widespread use of digital devices among children has raised concerns about the potential impact on their eye health. Excessive screen time can cause prolonged near focus, reduced outdoor time, and increased blue light exposure, all of which may contribute to myopia progression. Understanding the relationship between digital screen time and myopia progression is crucial for developing effective prevention and intervention strategies to mitigate the growing burden of myopia in children.

SUMMARY:
Research suggests that prolonged digital screen time is a significant contributing factor to the progression of myopia in children. Studies have shown that increased near-work activities, such as reading, writing, and screen time, can lead to an increased risk of developing myopia. The widespread use of digital devices among children has raised concerns about the potential impact on their eye health.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female myopic children of age 6 to 12 years were included with BCVA 6/6 with no any eye pathology.
* No medication or disease that could affect vision.
* Spherical equivalent of cylinder 0.50 to 1.00 were added.

Exclusion Criteria:

* Opacity, cataract, any fundus pathologies, strabismus or indication of previous ocular surgeries were excluded.
* High astigmatic children were excluded or more than 1.00DC.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Impact of Digital Screen Time in Progression of Myopia in Children he widespread use of digital devices among children has raised concerns about the potential impact on their eye health. Excessive screen time can cause prolonged near focus, reduced outdoor time, and increased blue light exposure, all of which may contribute to myopia progression.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
self admistred questioner | 12 Months
  self admistred questioner to check Mild, moderate, and severe Myopia in Children

CONTACTS AND LOCATIONS:
Locations (1):
- Watan optical, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No